CLINICAL TRIAL: NCT00009230
Title: Anti-Inflammatory Treatment for Age-Associated Memory Impairment: A Double-Blind Placebo-Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gary Small, MD, Professor of Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: IA0015; R01MH058156 (NIH); NCT00000185 (obsolete NCT alias)
Record Dates: First submitted 2001-01-23; First posted 2001-01-24 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Memory Disorders
Keywords: Age associated memory impairment; Mild cognitive impairment
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction | interventions — Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
This project is designed to study whether anti-inflammatory drugs, such as celecoxib, may delay age-related mental decline. We are also looking at genetic risk and brain structure as potential predictors of mental decline. We believe people with age-associated memory impairment who take celecoxib will show less evidence of mental decline than those receiving placebo (an inactive pill) after 18 months. We expect that brain structure at the start of the study, memory performance as indicated by tests, and age will be additional predictors of mental decline. We also predict that cognitive decline (i.e., decline in thinking and memory) and treatment response will vary according to genetic factors that may correlate with the age at which dementia begins. We believe other variables such as prior educational achievement, memory capability at the outset of the study, and gender may influence mental decline and treatment response. We will study people with age-associated memory impairment (mild memory complaints, decreased performance in selected memory tests), between 40 and 90 years of age. The subjects will be randomly (i.e., by a process similar to flipping a coin) assigned to treatment groups. The subjects will receive either an inactive substance (placebo) or celecoxib (400 mg/day). The subjects will receive a magnetic resonance imaging (MRI) scan, FDG PET scan, routine laboratory blood tests, electrocardiogram and cognitive tests. They will be followed for approximately 18 months and asked to return at specific intervals for follow-up testing. Measures of brain structure will be derived from baseline MRI scans and metabolic activity from PET scans, and blood will be drawn and tested to determine which forms (genotypes) of certain genetically determined cellular components the patient has.

DETAILED DESCRIPTION:
Several observational epidemiological studies indicate that anti-inflammatory treatments attenuate or prevent the symptoms of one of the most common mental disorders of late life, Alzheimer's disease (AD). Neuropathological studies also support inflammatory or immune mechanisms in AD, including findings of reactive microglia within or near AD lesions. Such evidence, however, is circumstantial, and controlled, randomized drug trials are needed to determine efficacy.

This project is designed to determine if the commonly used nonsteroidal anti-inflammatory drug (NSAID), celecoxib, is efficacious in delaying progression of cognitive symptoms in people with age-related cognitive losses who are at risk for developing AD. A total of 135 subjects with age-associated memory impairment (AAMI) who are at risk for further cognitive decline (age 40 to 90 years) will be randomized (double-blind design) to one of two treatment groups: celecoxib (400 mg/d) or placebo, and followed for 18 months. All randomized subjects will receive magnetic resonance imaging (MRI) scans, FDG PET scans, and selective genotyping (apolipoprotein E [APOE] and genetic risk for AD onset (e.g., APOE-4). Subjects receiving celecoxib are expected to show less evidence of cognitive decline than those receiving placebo. The proposed project builds upon our group's prior work on early detection of AD using brain imaging, genetic risk, and neuropsychological assessments. This project also is a logical follow-up to recent observational studies of a promising early intervention and will represent one of the first controlled, anti-inflammatory treatment trials for persons at high risk for age-related cognitive decline and the eventual development of AD.

Subjects will be followed closely to ensure that medication is safely used, without side effects (e.g., gastrointestinal, renal, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Age-associated memory impairment (AAMI)

Exclusion Criteria:

* Use of cholinesterase inhibitors
* Any current major psychiatric disorder such as depression or mania
* Subjects who may be sensitive to potential side effects of celecoxib, including those with any evidence of renal disease or gastrointestinal disease or predisposition or risk for bleeding, particularly gastrointestinal
* Subjects with histories of congestive heart failure, hypertension, peptic ulcer disease, any bleeding disorder, or other medical conditions that might increase medical risks from NSAID sensitivity
* Current diagnosis or history of alcoholism or drug dependence
* Evidence of depression
* Subjects with a contraindication for MRI scan
* Sulfur allergy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06 (Actual); Primary Completion 2005-06 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary W. Small, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Neuropsychiatric Institute, Los Angeles, California, United States